CLINICAL TRIAL: NCT01249157
Title: Histologic Assessment of the Difference Between 18F-2-fluoro-2-deoxy_D-glucose Positron Emission Mammography(PEM) and Magnetic Resonance Imaging (MRI) of the Breast
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10-189
Record Dates: First submitted 2010-11-24; First posted 2010-11-29 (Estimated); Results first posted 2015-12-24 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer
Keywords: MRI; PEM; 10-189
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Imaging

ARMS (1):
- MRI and PEM scans (Experimental): All consenting patients who are to have staging breast MRI, will be offered 18FDG PEM (Positron Emission Mammography) within 30 days. If the patient had a previous breast MRI that was done within 30 days at an outside institution, this MRI can be used if a radiologist determines that it is an adequate study. The surgery date will not be affected by the additional PEM evaluation. All imaging will be done and reviewed by MSKCC breast imagers. MRI and PEM findings suggestive of malignancy will be prospectively recorded in both the ipsilateral and contralateral breast.
  Interventions: Device: Positron Emission Mammography (PEM) and Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Device: Positron Emission Mammography (PEM) and Magnetic Resonance Imaging (MRI) — An additional 5 women will be enrolled at the beginning of the study for training purposes only and will not be included in the assessment of this study. Once the patient has had both breast MRI and PEM, the location of each site of potential breast cancer will be listed for each modality. The location of each abnormality on each imaging examination will be documented. Once the histopathologic evaluation has been performed, the pathology results will be compared to the imaging results for each modality. Furthermore, comparison of the performance of MRI and PEM will then be made with the pathological results as the truth. Comparison of the histology and biomarkers in each lesion detected by each modality will be done in order to determine if these factors affect detection by each modality.

SUMMARY:
Positron Emission Mammography (PEM) is a newly developed imaging examination of the breast that uses a radioactive glucose based tracer, which is a form of sugar attached to a low radiation agent, to detect cancer cells. The radioactive glucose based tracer is called fluorodeoxyglucose (FDG), and it is FDA approved. A PEM scanner is able to better detect cancer cells within the breast, more than a regular PET scanner. The PEM scanner is also FDA approved. This type of imaging may be able to see the breast cancer before it could be seen with mammograms and may be as good as or better than breast MRI.

The purpose of this study is to compare the value of FDG Positron Emission Mammography (PEM) with contrast enhanced Magnetic Resonance Imaging (MRI) of the breast for patients with breast cancer. This study will also perform special pathology test to compare the FDG PEM and contrast enhanced breast MRI images with the results from the standard of care breast surgery. This may teach us more about the biology of each breast tumor.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with recently diagnosed invasive or in situ breast cancer by core needle biopsy or FNA (confirmed at MSKCC) prior to enrollment.
* Patients planning treatment with mastectomy at MSKCC.
* Patients 21 years old or older.
* Patients who had or are having a breast MRI within 30 days or less of PEM.
* Patients who had or are having a digital mammogram.

Exclusion Criteria:

* Patients who are pregnant or breast feeding.
* Patients with prior radiation therapy or endocrine therapy.
* Patients who had a prior lumpectomy.
* Patients who are diabetic.
* Patients with moderate to end stage kidney disease.
* Patients who have a contraindication to MRI (i.e. pacemaker, metallic implants, etc).

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maxine Jochelson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Preoperative 18FDG PEM and MRI: Female patients with recently diagnosed invasive or in situ breast cancer
Period: Overall Study
Arm/Group | Preoperative 18FDG PEM and MRI
Started | 1
Completed | 0 (No data displayed because Outcome Measure has zero total participants analyzed.)
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The first 5 patients who consent to the study will be intended for training purposes only.
Groups:
- Preoperative 18FDG PEM and MRI: Female patients with recently diagnosed invasive or in situ breast cancer.The first 5 patients who consent to the study will be intended for training purposes only.
Arm/Group | Preoperative 18FDG PEM and MRI
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Accuracy of Preoperative 18FDG PEM
Description: using pathology as the gold standard and descriptively compare it to the accuracy of breast MRI in an exploratory analysis which will generate data for future studies. The first 5 patients who consent to the study were used for training purposes only.
Time Frame: 2 years
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Preoperative 18FDG PEM and MRI
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Preoperative 18FDG PEM and MRI
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The first 5 patients who consent to the study were used for training purposes only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes